CLINICAL TRIAL: NCT04336163
Title: Skin Imaging to Inform Laser Treatments
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: All 55 subjects enrolled in the study completed the initial study procedures, but due to the pandemic and the prolonged period where we were unable to follow up patients, we were not able to complete the aims for this protocol.
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Kristen Kelly, Professor of Dermatology, University of California, Irvine
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20195222
Record Dates: First submitted 2020-03-18; First posted 2020-04-07 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2023-11

CONDITIONS: Port-Wine Stain; Rosacea; Telangiectasia; Angioma
Keywords: Optical Coherence Tomography; Pulsed Dye Laser; Port-Wine Stain; Rosacea; Telangiectasia; Angioma
MeSH Terms: conditions — Port-Wine Stain; Rosacea; Telangiectasis; Hemangioma | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Intervention Model Description: A prospective study on the impact of Optical Coherence Tomography in laser treatment of vascular skin conditions.
Who Masked: Care Provider
Masking Description: For the control group, the laser surgeon would be unaware of OCT measurements of patients in the control group and would need to rely on his/her experience and intuition to determine the laser settings to treat the patient. For the experimental group, the laser surgeon will be exposed to the OCT measurements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Prospective Study Group (Experimental): For the experimental group, the laser surgeon will be exposed to the OCT measurements and will select laser settings and determine treatment parameters based on the measurements.
  Interventions: Device: Optical Coherence Tomography
- Prospective Control Group (Other): For the control group, the laser surgeon will not be exposed to the OCT measurements and will select laser settings and determine treatment parameters based on standard of care, intuition, and experience.
  Interventions: Device: Optical Coherence Tomography

INTERVENTIONS:
Device: Optical Coherence Tomography — Skin imaging to determine vascular characteristics such as plexus depth, vessel diameter, and vessel density.

SUMMARY:
The purpose of this study is to obtain information (such as lesion depth, depth of the most superficial part of the lesion, and the size and density of blood vessels) with the assistance of an imaging device, and use this information to assist in selection of laser settings for the treatment of skin conditions. The imaging modality is called Optical Coherence Tomography (OCT). Multiple laser modalities will be used, including intense pulsed light lasers (BroadBand Light, Profractional Sciton), pulsed dye lasers (Vbeam Perfecta, Candela), long-pulse 755nm lasers (GentleLASE, Candela), Sciton long-pulse 1064nm lasers, and non-ablative and ablative fractional resurfacing lasers (Profractional, Sciton). All of the lasers noted above are the only ones that will be used in this study. These lasers have 510k clearance and are being used as per their approved indications in this study. The choice of laser type is based on the skin lesion and is recommended by the physician, and the subjects who are going to enroll in this study will already be planned to undergo laser treatment as a standard of care for their condition. This is a pilot study that will explore the utility of skin imaging in guiding the laser treatment of skin lesions.

DETAILED DESCRIPTION:
The purpose of this research is to assist laser treatment of skin conditions by imaging the skin to obtain information about lesional skin. This is a pilot study that will explore the utility of skin imaging in guiding the laser treatment of skin lesions. This study will utilize Optical Coherence Tomography (OCT). Data acquisition of the skin will guide laser treatment by providing information on skin lesion characteristics.

There have been shown to be many applications for OCT. This imaging modality has been used to examine normal skin, burn scars, hemangiomas, nevus flammeus, fibrosarcomas, rosacea, and telangiectasias. Skin conditions to be studied include vascular lesions, scars, and inflammatory conditions. Normal and lesional skin will be assessed.

Currently, laser settings are selected without the assistance of imaging. Imaging with OCT provides more information about the characteristics of the skin lesion (such as lesion depth, depth of the most superficial part of the lesion, and the size and density of blood vessels), which could allow for more informed selection of laser settings to treat individual skin lesions. OCT has been used to examine laser treatments as well, but the proposed protocol would include the use of OCT to examine the stated skin lesions above before and after laser treatment in order to compare to historical/prospective controls that did not undergo OCT imaging. The goal of this study is to optimize laser treatment with the assistance of OCT and guide future laser treatments.

OCT is an imaging modality that uses light to image turbid media such as living tissues, and has been successfully used to generate high resolution (~10 micron) cross-sectional images of tissue microstructure in the human retina, skin, gastrointestinal tract, and genitourinary tract. OCT systems are now commercially available for ophthalmic and dermatologic use, and there are several clinical reports on the use of OCT in the vascular system and aero digestive tract, Ophthalmology, Pleural disorder, Neural tissue, Aneurysm healing, and Oral Pathology. This device focuses low power non-laser broad band infrared light onto tissue and does not involve input of significant amounts of energy into the subject; no temperature rise occurs. Because the wavelength of light used for imaging does not have adverse tissue effects, there is no risk.

Imaging with OCT provides information about the characteristics of the skin lesion (such as lesion depth, depth of the most superficial part of the lesion, and the size and density of blood vessels). OCT poses no known risks to the patients.

A multitude of studies have been conducted that validate the utility of OCT in imaging many types of skin lesions. Vascular lesions formulate a good portion of skin diseases studied by OCT, which includes rosacea, port-wine stain, hemangiomas, fibrosarcomas, cherry angiomas, and telangiectasias. Other studies have examined imaging of burn scars, the micro-circulation of the skin, and vascular changes with topical medical application. In all of these studies, OCT imaging aided treatment as well as provided a method to assess treatment outcome.

For port-wine stains, OCT has provided information such as vessel diameter and depth, which was discovered to be quite variable in port-wine stains, indicating that tailored laser treatments are likely to improve result. Byers et al. noted that OCT was a robust and non-invasive method for observing longitudinal dynamics of the subcutaneous microcirculation of tumors. Telangiectasias are a prominent feature of rosacea, and OCT has elucidated information about their treatment with intense-pulsed light to simply examine the effect of the treatment on the targeted lesions.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet the following inclusion criteria:

* Ability to understand and carry out subject instructions or be represented by a legally authorized guardian or representative.
* Ages 4 and older. Patients younger than 4 may have difficulty cooperating with the OCT measurements because each measurement requires the patient to remain still for approximately 30 seconds.
* Seeks and is scheduled for laser treatment of a skin lesion. Exclusion Criteria

Any of the following will exclude participation in the study:

* Inability to understand and/or carry out subject instructions.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen M Kelly, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No
All co-researchers and research personnel only on this IRB protocol will have access to IPD.

REFERENCES:
- [Result] Waibel JS, Holmes J, Rudnick A, Woods D, Kelly KM. Angiographic optical coherence tomography imaging of hemangiomas and port wine birthmarks. Lasers Surg Med. 2018 Mar 22. doi: 10.1002/lsm.22816. Online ahead of print. PMID 29566276
- [Result] Waibel JS, Rudnick AC, Wulkan AJ, Holmes JD. The Diagnostic Role of Optical Coherence Tomography (OCT) in Measuring the Depth of Burn and Traumatic Scars for More Accurate Laser Dosimetry: Pilot Study. J Drugs Dermatol. 2016 Nov 1;15(11):1375-1380. PMID 28095550
- [Result] Byers RA, Fisher M, Brown NJ, Tozer GM, Matcher SJ. Vascular patterning of subcutaneous mouse fibrosarcomas expressing individual VEGF isoforms can be differentiated using angiographic optical coherence tomography. Biomed Opt Express. 2017 Sep 19;8(10):4551-4567. doi: 10.1364/BOE.8.004551. eCollection 2017 Oct 1. PMID 29082084
- [Result] Aldahan AS, Chen LL, Tsatalis JP, Grichnik JM. Optical Coherence Tomography Visualization of a Port-Wine Stain in a Patient With Sturge-Weber Syndrome. Dermatol Surg. 2017 Jun;43(6):889-891. doi: 10.1097/DSS.0000000000001055. No abstract available. PMID 28541265
- [Result] Themstrup L, Ciardo S, Manfredi M, Ulrich M, Pellacani G, Welzel J, Jemec GB. In vivo, micro-morphological vascular changes induced by topical brimonidine studied by Dynamic optical coherence tomography. J Eur Acad Dermatol Venereol. 2016 Jun;30(6):974-9. doi: 10.1111/jdv.13596. Epub 2016 Feb 25. PMID 26916576
- [Result] Aldahan AS, Mlacker S, Shah VV, Chen LL, Nouri K, Grichnik JM. Utilization of Optical Coherence Tomography in the Evaluation of Cherry Hemangiomas. J Drugs Dermatol. 2016 Jun 1;15(6):713-4. PMID 27272077
- [Result] Themstrup L, Welzel J, Ciardo S, Kaestle R, Ulrich M, Holmes J, Whitehead R, Sattler EC, Kindermann N, Pellacani G, Jemec GB. Validation of Dynamic optical coherence tomography for non-invasive, in vivo microcirculation imaging of the skin. Microvasc Res. 2016 Sep;107:97-105. doi: 10.1016/j.mvr.2016.05.004. Epub 2016 May 25. PMID 27235002
- [Result] Urban J, Siripunvarapon AH, Meekings A, Kalowitz A, Markowitz O. Optical coherence tomography imaging of erythematotelangiectatic rosacea during treatment with brimonidine topical gel 0.33%: a potential method for treatment outcome assessment. J Drugs Dermatol. 2014 Jul;13(7):821-6. PMID 25007365
- [Result] Ring HC, Mogensen M, Banzhaf C, Themstrup L, Jemec GB. Optical coherence tomography imaging of telangiectasias during intense pulsed light treatment: a potential tool for rapid outcome assessment. Arch Dermatol Res. 2013 May;305(4):299-303. doi: 10.1007/s00403-013-1331-z. Epub 2013 Mar 2. PMID 23455486
- [Result] Mogensen M, Bojesen S, Israelsen NM, Maria M, Jensen M, Podoleanu A, Bang O, Haedersdal M. Two optical coherence tomography systems detect topical gold nanoshells in hair follicles, sweat ducts and measure epidermis. J Biophotonics. 2018 Sep;11(9):e201700348. doi: 10.1002/jbio.201700348. Epub 2018 Jun 19. PMID 29611306
- [Result] Banzhaf CA, Thaysen-Petersen D, Bay C, Philipsen PA, Mogensen M, Prow T, Haedersdal M. Fractional laser-assisted drug uptake: Impact of time-related topical application to achieve enhanced delivery. Lasers Surg Med. 2017 Apr;49(4):348-354. doi: 10.1002/lsm.22610. Epub 2016 Nov 25. PMID 27885682
- [Result] Olesen UH, Mogensen M, Haedersdal M. Vehicle type affects filling of fractional laser-ablated channels imaged by optical coherence tomography. Lasers Med Sci. 2017 Apr;32(3):679-684. doi: 10.1007/s10103-017-2168-z. Epub 2017 Feb 17. PMID 28213875

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prospective Study Group | Prospective Control Group
Started | 55 | 0
Completed | 0 | 0
Not Completed | 55 | 0
Not completed — Lost to Follow-up | 55 | 0

BASELINE CHARACTERISTICS:
Population: 55 experimental group subjects were consented to this study. However, due to the global pandemic, subjects could not come for study visits, which significantly precluded the study team from following up with the subjects for several months. Therefore, the study was terminated. The preoperative photographs could not be compared to the postoperative photographs since the subjects could not be followed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prospective Study Group | Prospective Control Group | Total
Number analyzed (Participants) | 55 | 0 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 |  | 8
  Between 18 and 65 years | 38 |  | 38
  >=65 years | 9 |  | 9
Age, Continuous [Mean (Full Range); unit: years] | 46 [4 to 89] |  | 46 [4 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 0 | 45
  Male | 10 | 0 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 15 |  | 15
  Unknown or Not Reported | 40 |  | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 40 | 0 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 0 | 7
Region of Enrollment [Number; unit: participants]
  United States | 55 |  | 55

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Change in Photographed Lesion
Description: Primary outcome variable includes assessment of change in photographed lesion. Two board-certified dermatologists will grade the degree of change of the photographed lesion in quartiles (no change or darkening=0-25, mild lightening=26-50, good lightening=51-75, excellent lightening=76-95, complete resolution=96-100).
Time Frame: Through study completion; average of one year
Population: 55 experimental group subjects were consented to this study. However, due to the global pandemic, subjects could not come for study visits, which significantly precluded the study team from following up with the subjects for several months. Therefore, the study was terminated. Although we have preoperative photographs, we did not have postoperative photographs of the subjects because we were not able to see them in followup.
Arm/Group | Prospective Study Group | Prospective Control Group
Number analyzed (Participants) | 0 | 0

2. Other Pre Specified Outcome: Number of Participants With Scarring, Blistering, Bruising, and Scabbing
Description: Any adverse effects of treatment such as scarring, blistering, bruising, and scabbing.
Time Frame: Through study completion; average of one year
Population: 55 experimental group subjects were consented to this study. However, due to the global pandemic, subjects could not come for study visits, which significantly precluded the study team from following up with the subjects for several months. Therefore, the study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Study Group | Prospective Control Group
Number analyzed (Participants) | 55 | 0
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline to study completion, on average 1 year.
Description: Number of subjects at risk for adverse events is 55. 55 experimental group subjects were consented to this study. However, due to the global pandemic, subjects could not come for study visits, which significantly precluded the study team from following up with the subjects for several months. Therefore, the study was terminated.
Arm/Group | Prospective Study Group | Prospective Control Group
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/0
Other Adverse Events (participants affected / at risk) | 0/55 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT04336163/Prot_SAP_ICF_002.pdf